CLINICAL TRIAL: NCT01007422
Title: Opioid Titration In the Hospice Setting: Barriers Assessment and Modification of the Model Order Sheet and Protocol Stage 2, Part B
Brief Title: Opioids Titration in Hospice Patients
Status: Withdrawn | Type: Observational
Why Stopped: Issues with Hospice
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine; Director, Cancer Supportive Care Program; Director, Head and Neck Research Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC SUPP 0822; P30CA068485 (NIH); VU-VICC-SUPP-0822; VU-VICC-IRB-IRB-080370
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Pain; Solid Tumor
Keywords: unspecified adult solid tumor, protocol specific; pain
MeSH Terms: conditions — Pain | interventions — Therapeutics; Analgesia; Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Supportive Care
  Interventions: Behavioral: telephone-based intervention; Other: communication intervention; Other: intervention by caregiver; Other: medical chart review; Other: survey administration; Procedure: end-of-life treatment/management; Procedure: pain therapy; Procedure: psychosocial assessment and care

INTERVENTIONS:
Behavioral: telephone-based intervention
Other: communication intervention
Other: intervention by caregiver
Other: medical chart review
Other: survey administration
Procedure: end-of-life treatment/management
Procedure: pain therapy
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Opioids lessen pain caused by cancer. Titration of opioids in the hospice setting is suboptimal due to numerous barriers. Order sets may help to provide timely and effective medical and pharmaceutical intervention.

PURPOSE: The purpose of this study was to identify barriers to good pain control in the hospice setting and to develop an order set that would safely address these barriers.

DETAILED DESCRIPTION:
Objective 1:

To assess barriers to pain control in the hospice setting.

Using a mixed methods approach, key stakeholders including physicians, nurses, patients and caregivers were queried about pain control in the hospice setting, barriers to pain control and the desirability of an order set to address this issue.

Objective 2:

To develop and conduct pilot testing of an order set designed to improve pain control in the hospice setting.

An opioid titration order sheet based on our previous R0-1 was modified based on the information derived from the interviews and questionnaires completed by the physicians, nurses, patients and caregivers.

A cohort of 20 patients were enrolled on the first phase of the pilot study in order to test the modified pain assessment form and the feasibility administration of the study materials to be completed by the patient and caregiver. Forms are as follows:

* Patient assessment: At baseline, patients provide demographic data and complete the Pain Assessment Form and the Pain Communication Survey. The pain assessment form addresses average pain, worst pain, pain relief, hours in pain, pain-related distress, and barriers to pain control. Patients are asked to rate pain control. Patients also complete the Pain Communication Survey to assess how they communicate with healthcare providers about their pain. After the baseline assessment is completed, patients complete the Pain Assessment form on a daily basis. Pain is also assessed by the research nurse at least 3 times weekly (1 home visit* and 2 telephone interviews). Patients are followed until the time of death.

NOTE: *If a patient is hospitalized or transferred to the inpatient hospice facility, the patient interview will take place there.

* Caregiver assessment: At baseline, caregivers complete a demographic survey, a Pain Assessment Form, the Pain Communication Survey, Caregiver Self-Efficacy in Pain Management Scale (CSEPMS), Caregiver Pain Management Questionnaire (CPMQ), and the Stressful Caregiver Adult Reactions to Experiences of Dying (SCARED). Caregivers are then interviewed by the study nurse using the Pain Assessment Form as a guideline to obtain more detailed information about adequacy of the patient's pain control, side effects of medication, barriers to pain control, and caregiver concerns and burden. Follow-up data from caregivers is obtained through completion of CSEPMS, CPMQ, and SCARED questionnaires and their assessment of patient's pain form at the end of weeks 1, 2, and 3.
* Chart review: A research nurse conducts a chart review after patient's death. Cancer and cancer-related treatment data is obtained and documentation about pain management is recorded. From the time of study entry, all staff notes are reviewed to document pain assessment, calls to physician or other support personnel (including pharmacy calls), identified barriers to pain control, and treatment modifications (including medications to treat side effects).

After 20 patients, it was deemed not feasible to complete the study forms and to recruit adequately for the trial. The study was suspended.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Outpatient at the Alive Hospice in the State of Tennessee

    * Diagnosed with carcinoma
    * Pain requiring fixed-dose opioids
  * Caregiver for an Alive Hospice patient

    * Any caregiver who is identified by the patient is eligible

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Able to speak/comprehend English
* Lives within a 60-mile radius of Alive Hospice

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out-patient hospice patients.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To obtain determine the safety and feasibility of an opioid titration order sheet in the hospice setting. | at 4 weeks
  Pain assessments will be completed at baseline and daily for 4 weeks. Survey instruments will be completed at the end of weeks 1, 2, and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Murphy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center